CLINICAL TRIAL: NCT03976141
Title: Validation of a New Topographic Classification of Bone Marrow Lesions of the Knee
Brief Title: New Topographic Classification of Knee Bone Marrow Lesions
Acronym: ncbe
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Pietro Randelli, MD, Professor, University of Milan
Other Study IDs: ncbe
Record Dates: First submitted 2019-05-17; First posted 2019-06-05 (Actual); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Knee Bone Marrow Lesions
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- a
  Interventions: Diagnostic Test: mri

INTERVENTIONS:
Diagnostic Test: mri — knee mri

SUMMARY:
the investigator are studying a new topographic classification of bone marrow lesion in the knee and validating it.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 with mri with lesion consent given

Exclusion Criteria:

* under mri previous surgery tumors no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: exam in 2018
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The researchers will calculate the prevalence of BMLs in knee MRI and calculate the intra-observer and inter-observer reliability of the new classification proposed. | The lesions will be evaluated on knee MRI performed in the period between January 2017 to December 2018
  This study proposes a topographic classification for knee BMLs consisting in 5 different types of lesions. the classification proposed will be validated by 3 independent researchers.

CONTACTS AND LOCATIONS:
Locations (1):
- 2) 1° Clinica Ortopedica, ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO, Milan, Milan, Italy